CLINICAL TRIAL: NCT02167230
Title: Effect of Jailed-Balloon Technique in Percutaneous Coronary Intervention for Non-Left Main Coronary Bifurcation Lesions: A Prospective, Randomized Study.
Brief Title: Jailed-balloon Technique in Coronary Bifurcation Lesion PCI
Acronym: JBTinCBL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guangdong Provincial People's Hospital (Other)
Collaborators: Shenzhen People's Hospital (Other); Kashgar 1st People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JBT
Record Dates: First submitted 2014-06-17; First posted 2014-06-19 (Estimated); Last update posted 2014-06-19 (Estimated); Status verified 2014-06

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Artery Disease; Percutaneous Coronary Intervention; Bifurcation; Jailed-balloon technique
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Jailed-balloon technique (Experimental): Apply jailed-balloon technique to protect the side branch during coronary bifurcation PCI
  Interventions: Procedure: Jailed-balloon technique
- Jailed-wire technique (Active Comparator): Apply jailed-wire technique to protect the side branch during coronary bifurcation PCI
  Interventions: Procedure: Jailed-wire technique

INTERVENTIONS:
Procedure: Jailed-balloon technique — A monorail balloon is placed in the side branch(SB) before the stent in main branch(MB) is deployed. After MB stent is deployed to nominal pressure, the balloon in SB is inflated to 3 atm generally but to higher pressure to perform angioplasty if the blood flow in SB is compromised. The balloon in SB is then removed while the wire in SB is left in place. The MB stent balloon is inflated again for stent apposition. The SB wire is left in place to facilitate rewiring if the blood flow in SB is compromised. Otherwise the SB wire is removed after the stent balloon is inflated again.
  Arms: Jailed-balloon technique
Procedure: Jailed-wire technique — A percutaneous transluminal coronary angioplasty(PTCA) wire is placed in the side branch(SB) before the stent in main branch(MB) is deployed. After MB stent is deployed to some pressure to achieve full apposition, the wire in SB is left in place to facilitate rewiring if the blood flow in SB is compromised. Otherwise the SB wire is removed after the MB stent is deployed.
  Arms: Jailed-wire technique

SUMMARY:
This study aims to test the hypothesis that jailed-balloon technique(JBT) is superior to jailed-wire technique(JWT) in non-left main coronary bifurcation percutaneous coronary intervention(PCI) by lowering the risk of side branch(SB) loss and PCI related myocardial infarction, as well as 1-year major adverse cardiovascular events(MACEs).

DETAILED DESCRIPTION:
1. Objective: To compare the protective effect between JBT and JWT during PCI for non-left main coronary bifurcation lesions.
2. Background: Solid evidence is scant to compare the protective effect between JBT and JWT during PCI for non-left main coronary bifurcation lesions.
3. Study design: This is a multi-center, prospective, randomized study.
4. Methods

4a. Study populations: Patients with non-left main coronary bifurcation lesions(Medina 1,1,1 ), which SBs are less than 2.5mm and more than 1mm, are enrolled in this study. Patients are randomized to JBT group and JWT group.

4b. Procedure: For patients enrolled in JBT group, a monorail balloon is placed at the ostium of SB to protect the SB before the stent in main branch(MB) is deployed. Only a PTCA wire would be placed in the SB while stenting MB for patients randomized in JWT group. Only drug-eluting stent should be implanted in the target vessel.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years and ≤75 years;
2. De novo Medina 1,1,1 coronary bifurcation with a main branch(MB) >2.5mm while side branch <2.5mm and >1.5mm;
3. Only one bifurcation lesion need to be treated in one vessel;
4. The target lesion in MB has stenosis more than 75% or fractional flow reserve(FFR) less than 0.75 and the stenosis in SB ostium is more than 50%;
5. Signed consent is obtained.

Exclusion Criteria:

1. Left ventricular ejection fraction(LVEF) less than 30%;
2. Hemodynamic instability or cardiac shock;
3. Myopathy or muscular injury with elevation of creatine kinase to more than 3mg/dL;
4. Tumor with expected survival less than 1 year;
5. Autoimmune disease;
6. Active gastrointestinal bleeding or any contraindication for dual antiplatelet therapy;
7. Acute coronary syndrome require emergency PCI;
8. Coronary bifurcation need to be treated with two-stent strategy;
9. Not suitable for drug-eluting stent(DES) implantation;
10. Mental disorder or alcohol dependence;
11. PCI or coronary artery bypass graft (CABG) within 6 months before enrollment;
12. Target lesion is in-stent restenosis;
13. Women in gestation period or lactation period or human chorionic gonadotropin (HCG) urine test positive.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 410 (Estimated)
Dates: Start 2014-10; Primary Completion 2016-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Side branch(SB) loss and PCI related myocardial infarction | Within 48 hours after PCI
  The primary outcome of the study is a composite of SB loss or PCI related myocardial infarction.
  According to Thrombolysis in Myocardial Infarction (TIMI) flow grading system, SB loss is defined as less than TIMI 3 flow immediately following MB stenting. It is considered temporary SB loss if TIMI 3 flow is restored with angioplasty and/or stenting. Otherwise, SB loss is considered permanent.
  In patients with normal (≤99th percentile URL) baseline cardiac troponin(cTn) concentrations, PCI related myocardial infarction is defined as elevations of cTn >5× 99th percentile URL occurring within 48 hours of the procedure, which should be accompanied with other evidence of myocardial injury. A rise of >20% is required for the diagnosis of PCI related myocardial infarction if the baseline cTn values are elevated and are stable or falling.

SECONDARY OUTCOMES:
Major adverse cardiovascular events(MACEs) | Within 1 year after PCI
  MACEs is a composite end point including cardiac death, non fatal myocardial infarction and target vessel revascularization(TVR).
PCI related complication | Immediately after PCI
  PCI related complication include coronary dissection, coronary perforation, device dislodgement, device entrapment and device rupture.

CONTACTS AND LOCATIONS:
Overall Officials: Jiyan Chen, Doctor, Study Chair — Guangdong Provincial People's Hospital; Jianfang Luo, Doctor, Study Director — Guangdong Provincial People's Hospital; Pengcheng He, Doctor, Principal Investigator — Guangdong Provincial People's Hospital
Locations (2):
- China (2):
  - Shenzhen People's Hospital, Shenzhen, Guangdong
  - Kashgar District 1st People's Hospital, Kashgar, Xinjiang

REFERENCES:
- [Background] Sharma SK, Sweeny J, Kini AS. Coronary bifurcation lesions: a current update. Cardiol Clin. 2010 Feb;28(1):55-70. doi: 10.1016/j.ccl.2009.10.001. PMID 19962049
- [Background] Latib A, Colombo A. Bifurcation disease: what do we know, what should we do? JACC Cardiovasc Interv. 2008 Jun;1(3):218-26. doi: 10.1016/j.jcin.2007.12.008. PMID 19463303
- [Background] Depta JP, Patel Y, Patel JS, Novak E, Yeung M, Zajarias A, Kurz HI, Lasala JM, Bach RG, Singh J. Long-term clinical outcomes with the use of a modified provisional jailed-balloon stenting technique for the treatment of nonleft main coronary bifurcation lesions. Catheter Cardiovasc Interv. 2013 Nov 1;82(5):E637-46. doi: 10.1002/ccd.24778. Epub 2013 Jul 30. PMID 23420654
- [Background] Colombo F, Biondi-Zoccai G, Infantino V, Omede P, Moretti C, Sciuto F, Siliquini R, Chiado S, Trevi GP, Sheiban I. A long-term comparison of drug-eluting versus bare metal stents for the percutaneous treatment of coronary bifurcation lesions. Acta Cardiol. 2009 Oct;64(5):583-8. doi: 10.2143/AC.64.5.2042686. PMID 20058502
- [Background] Singh J, Patel Y, Depta JP, Mathews SJ, Cyrus T, Zajarias A, Kurz HI, Lasala JM, Bach RG. A modified provisional stenting approach to coronary bifurcation lesions: clinical application of the "jailed-balloon technique". J Interv Cardiol. 2012 Jun;25(3):289-96. doi: 10.1111/j.1540-8183.2011.00716.x. Epub 2012 Feb 26. PMID 22364484